CLINICAL TRIAL: NCT03634852
Title: A Two Different Chemoprophylaxis Approaches After Phacoemulsification Surgery in One Thousand Patients in Iraq :a Clinical Trial
Brief Title: A Two Chemoprophylaxis Approaches After Phacoemulsification Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Suzan A Rattan (Other)
Collaborators: Al-Kindy College of Medicine (Other)
Responsible Party: Sponsor-Investigator, Suzan A Rattan, Assistant professor in ophthalmology, Al-Kindy College of Medicine
Organization: Al-Kindy College of Medicine (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2 Al-KindyCM
Record Dates: First submitted 2018-07-31; First posted 2018-08-17 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2018-08

CONDITIONS: Endophthalmitis Postoperative
Keywords: IC Moxifloxacin hydrochloride; SC triamcinolone acetonide
MeSH Terms: interventions — Moxifloxacin; Ophthalmic Solutions; Dexamethasone

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Topical (Active Comparator): Moxifloxacin hydrochloride 0.5% eye drops and dexamethasone 0.1% eye drops were prescribed four times a day for 1 month postoperatively.
  Interventions: Drug: Moxifloxacin hydrochloride 0.5% eye drops; Drug: Dexamethasone 0.1% eye drops
- Intracameral - Subconjunctival (Active Comparator): Intracameral Moxifloxacin 0.1% with Subconjunctival Triamcinolone acetonide 4 mg /0.4 ml had been administered at the conclusion of the surgery
  Interventions: Drug: Intracameral Moxifloxacin 0.1%; Drug: Subconjunctival Triamcinolone acetonide 4 mg /0.4 ml

INTERVENTIONS:
Drug: Moxifloxacin hydrochloride 0.5% eye drops — were prescribed four times a day for 1-month postoperatively
  Other Names: Vigamox eye drops
  Arms: Topical
Drug: Dexamethasone 0.1% eye drops — were prescribed four times a day for 1-month postoperatively
  Other Names: Maxidex eye drops
  Arms: Topical
Drug: Intracameral Moxifloxacin 0.1% — Auromox (0.5%): is a sterile clear yellow pale colored preservative free isotonic ophthalmic solution with pH 6.0 to 7.5 and osmolarity 620 -320 milliosmol ( mOsm).The sterile Auromox vial contains 1cc Moxifloxacin hydrochloride 5.45 mg equivalent to 5mg of Moxifloxacin. This product is manufactured by Aurolab an Indian pharmaceutical company. Auromox is available in many countries including Iraq.
  Each vial enough for 15 different patients by using a sterile needle and 5cc syringe. By the sterile hand's, the surgeon draws the whole 1cc of Moxifloxacin 0.5% and diluted with 4 cc of balanced salt solution (BSS) to get 5 mg in 5 cc (0.1%) then draw 0.2 cc for each patient.
  Other Names: Auromox
  Arms: Intracameral - Subconjunctival
Drug: Subconjunctival Triamcinolone acetonide 4 mg /0.4 ml — Aurocort is a preservative-free Triamcinolone acetonide (40 mg /1cc), with along acting depot preparation of triamcinolone in 1cc vial also the product of Aurolab company and commercially available in our country.
  The whole 1cc had been drawn and diluted with 3cc of BSS and SC injection of 4 mg in 0.4 cc of Triamcinolone was given (as a final step in the surgery) 6mm from the limbus usually an inferotemporal site that is easily accessible and the plaque that formed will be not visible within palpebral fissure
  Other Names: Aurocort
  Arms: Intracameral - Subconjunctival

SUMMARY:
Post cataract surgery bacterial endophthalmitis is a rare but the most devastating complication with a poor visual outcome.

The preferred pattern of chemoprophylaxis varied world widely. The use of preoperative povidone iodine is universal. Most European surgeons prefer the use of Intracameral (IC) antibiotics whereas topical fluoroquinolone that prescribed perioperatively is the most common pattern in the United state(US). The current study aimed to evaluate the effectivity and safety of a combination of diluted IC Moxifloxacin and subconjunctival (SC) Triamcinolone acetonide as prophylaxis of bacterial endophthalmitis and postoperative inflammation in five hundred phacoemulsification surgeries and compare its results with the same number of patients treated by topical Moxifloxacin hydrochloride and Dexamethasone eye drops when given four times a day for 1month postoperatively.

DETAILED DESCRIPTION:
Study design and populations:

The current clinical trial included a total 1000 patients with visually significant cataract scheduled to have phacoemulsification surgery at an Eye specialty private hospital in Baghdad /Iraq during 18 months period from 1st of October 2016 to 1st of February 2018 by two surgeons.

The current two methods of prophylaxis of postoperative endophthalmitis and inflammation were discussed with the patients and informed consent was obtained about the treatment and the enrollment in the current study.

Two methods of prophylaxis of postoperative bacterial endophthalmitis and inflammation were planned to use. For 500 patients (group 1) topical moxifloxacin hydrochloride 0.5% (Vigamox,Alcon) and dexamethasone 0.1%(Maxidex, Alcon) eye drops prescribed four times a day for 1-month postoperatively ,while for the remaining 500 patients (group 2), intracameral (IC) diluted moxifloxacin 0.1% and subconjunctival triamcinolone acetonide 4 mg/0.4 cc is the combination that planned to used for prophylaxis.

Preoperative evaluations:

The two surgeons follow the same protocol for the preoperative evaluation including slit lamp, Goldmann applanation tonometry(AT900, Haag-Streit Diagnostics, Switzerland), dilated fundus examination and macular optical coherence tomography (OCT)(Optovue, RTVue-100, Fremont, CA).

Follow- up visits were on the first postoperative day, 1week, 1 month, and 3months postoperatively.

The mean age of patients in group 1 was 59.4 years ± 9.04, 300 were female and 200 were male, 160 with type 2 diabetes mellitus without retinopathy and the preoperative intraocular pressure (IOP) range were from 10 to 25 mmHg with mean 14.49 mmHg ± 3.11.

Group 2 patients had a mean age of 59.7 ±8.84, 320 were female and 180 were male, 140 with good controlled diabetes and preoperative IOP mean was 14.47 mmHg ±3.10 range was from 9.5-20.6 mmHg.

statistical analysis: Minitab 16 software used for data statistical analysis, data were expressed in mean ± standard deviation (SD), for each group the preoperative baseline versus the corresponding postoperative data were compared by paired-sample t-test, while for the comparison of the 2 independent groups we used two-sample t-test and the results considered statistically significant if P value < 0.05.

ELIGIBILITY:
Inclusion Criteria: for both groups; the patients with visually significant cataract were included in the current study should have

1. no current or previous intraocular inflammation,
2. no history of glaucoma or topical corticosteroid responsiveness.
3. All the included patients had normal preoperative fundus examination and normal preoperative macular OCT.
4. All the patients who have the above-mentioned inclusion criteria were included in the current comparison whether phacoemulsification surgery was complicated or not.

Exclusion Criteria:

1. For group 2; any patient used a topical antibiotic, nonsteroidal anti-inflammatory drug (NSAID) or corticosteroid up to 1 week before the planned day of surgery,
2. any patient with a history of glaucoma or steroid responsiveness
3. any patient with significant maculopathy were excluded from the current comparison.

Ages: 38 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Actual)
Dates: Start 2016-10-01 (Actual); Primary Completion 2018-02-01 (Actual); Study Completion 2018-02-01 (Actual)

PRIMARY OUTCOMES:
Incidence of Bacterial endophthalmitis in 1000 phacoemulsification surgeries | The duration of follow up for each patient was a 3 months postoperatively.
  All patients assessed by slit lamp examination for possibility of early or late onset bacterial endophthalmitis after phacoemulsification surgery.

SECONDARY OUTCOMES:
Intraocular pressure(IOP) was measured on 1week,1month,and 3 months visits by Goldmann applanation tonometry . | The duration of follow up for each patient was a 3 months postoperatively.
  For all patients IOP was measured during the last 3 visits to exclude the possibility of significant IOP elevation (> 10 mmHg from the base line) after phacoemulsification surgery with the use of 2 different methods of chemoprophylaxis and to show which of them has the more possibility to increase IOP

OTHER OUTCOMES:
Break through inflammation (A significant anterior chamber reaction that may notice after 10 days postoperatively). | The duration of follow up for each patient was a 3 months postoperatively.
  The anterior chamber(AC ) reaction was estimated by slit lamp and the grading had been done according to the Standardization of Uveitis Nomenclature (SUN) Working Group,all patients assessed for possibility of significant sterile intraocular inflammation after 10 days postoperatively.
Central macular thickness (CMT) | OCT was done preoperatively and 3 months postoperatively.
  Macular optical coherence tomography (OCT) was done preoperatively and 3 months postoperatively for all patients to show the possibility of increased macular thickness after phacoemulsification surgery with the use of different chemoprophylaxis methods.

IPD SHARING:
Plan to Share IPD: No